CLINICAL TRIAL: NCT06484244
Title: Locomotion Adaptation Deficits in Older Adults With Mild Cognitive Impairment and Alzheimers Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Trisha Kesar, Associate Professor, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00006698; R21AG084231 (NIH)
Record Dates: First submitted 2024-06-26; First posted 2024-07-03 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Alzheimers Disease; Mild Cognitive Impairment
Keywords: walking function; gait disturbances; gait variability; locomotor adaptation
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Mobility Limitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Split-beltTreadmill-based Locomotor Adaptation in Older Adults with MCI (Experimental): Older adults with mild cognitive impairment (MCI) complete 5 split-belt treadmill walking exercise sessions over a 2-week period.
  Interventions: Other: 5 Sessions of Split-belt Treadmill-based Locomotor Adaptation
- Split-beltTreadmill-based Locomotor Adaptation in Older Adults with AD (Experimental): Older adults with Alzheimer's Disease (AD) complete 5 split-belt treadmill walking exercise sessions over a 2-week period.
  Interventions: Other: 5 Sessions of Split-belt Treadmill-based Locomotor Adaptation

INTERVENTIONS:
Other: 5 Sessions of Split-belt Treadmill-based Locomotor Adaptation — Participants will complete 5 sessions of split-belt treadmill-based locomotor adaptation. The split-belt instrumented treadmill allows the two belt speeds to be operated independently, enabling different belt speeds for each leg. The split-belt walking assessment will consist of 3 phases: baseline phase in which the belts operated at the same speed (Pre-tied, 2-minutes), a phase in which the belts operated at different speeds (Split-belt, 15-minutes), and a final phase in which the belts operated at the same speed (Post-tied, 4-minutes).

SUMMARY:
In people with Mild Cognitive Impairment (MCI) and Alzheimer's Disease (AD), reduced capacity for locomotor adaptation is a fundamental but poorly understood mechanism that can be a sensitive biomarker of cognitive-motor impairments. It is also an important therapeutic target for exercise-based interventions to improve walking function. The overall goal of this study is to understand the effects of MCI and AD on locomotor adaptation and walking function.

DETAILED DESCRIPTION:
In conjunction with cognitive impairments, older adults with Alzheimer's Disease (AD) and Mild Cognitive Impairment (MCI) show increased impairments in walking function throughout disease progression. The ability to walk without the risk of falling is necessary for independent community activity and participation for elderly individuals. However, the relationships between cognition, gait dysfunction, and fall risk in people with MCI and AD are poorly understood, warranting further study. The objective of this study is to test the researchers' central hypothesis that in people with MCI and AD, decreased capacity for locomotor adaptation can worsen disease progression, and lead to reduced motor-cognitive function, mobility, and quality of life.

Community-based walking function requires complex motor coordination, sensory feedback, dynamic balance, adaptation to changing environmental stimuli, while also engaging in attentional tasks such as crossing a busy street or talking over the phone. Unfortunately, cognitive dysfunction, the hallmark of MCI and AD, directly impacts the cognitive-motor neural resources needed to carry out activities of daily living. People with MCI and AD walk slower, fall more, and have deficits in gait performance variables such as stride symmetry, and step regularity. Importantly, gait disturbances have often been shown to precede cognitive decline. In this study, the researchers propose to test their hypothesis that a decline in locomotor adaptation capacity may explain gait and mobility deficits in people with MCI and AD. Locomotor adaptation is a fundamentally important process that enables humans to flexibility respond to environmental demands, enabling normal community walking function. Split-belt adaptation is a standardized, robust, well studied paradigm for quantifying a person's capacity for locomotor adaptation, but had not yet been evaluated in people with MCI and AD. Split-belt walking task assesses locomotor adaptation, i.e. the ability to adjust stepping movements to changing environmental demands via trial-and-error processing. The split-belt task is systematically assessed during treadmill walking, where the speed of each leg can be controlled independently such that one belt and the corresponding leg run at a different speed (e.g., twice as fast or a 2:1 speed ratio) than the other leg. In previous work, both the magnitude and rate of split-belt adaptation as well as de-adaptation (during the after-effect) have provided objective measures of an individual's locomotor adaptation capacity.

The researchers of this study hypothesize that decreased capacity for split-belt adaptation may be an important contributing factor and a potentially sensitive indicator of increased fall risk and cognitive decline in older individuals with MCI and AD.

The researchers will examine locomotor adaptation capacity with three study aims: Aims 1 and 2 are observational, assessing walking function among persons with MCI and AD and age-matched controls. In Aim 3, a clinical trial is performed to evaluate the feasibility of a split-belt walking intervention on walking function in older adults with MCI and AD. Ten participants (5 with MCI and 5 with AD) will complete 5 split-belt treadmill walking exercise sessions over a 2-week period. The primary and secondary outcome measures for this study are measured in evaluation sessions before (Pre-training) and after 5 training sessions (Post-training).

ELIGIBILITY:
Inclusion Criteria:

* AD and MCI will be defined through formal diagnosis provided by a board-certified Neurologist. Amnestic MCI will be defined using the AD Neuroimaging Initiative (ADNI) criteria. All MCI participants in ADNI are required to have an amnestic subtype defined as:

  * Subjective memory concern or a memory problem noted by their partner
  * Abnormal memory function documented by a specified education adjusted cutoff score on the delayed paragraph recall of the Anna Thompson story of the Logical Memory subtest from the Wechsler Memory Scale-Revised
  * Mini-Mental State Exam (MMSE) score between 20 and 26 (inclusive). Exceptions may be made for subjects with less than 8 years of education at the discretion of the PI. (iv) Single or multi-domain amnestic MCI (both subtypes are at high risk for progression to AD)
  * Clinical Dementia Rating (CDR) = 0.5 (Memory Box score must be at least 0.5)
  * General functional performance sufficiently preserved
* Evidence of impaired executive function based on Montreal Cognitive Assessment (MoCA) score 13-17
* Able to walk 10 or more feet without an assistive device
* Completed six grades of education or has a good work history (sufficient to exclude intellectual disabilities)
* Not hospitalized within the last 60 days

Exclusion Criteria:

* Acute medical illness requiring hospitalization
* Uncontrolled congestive heart failure
* History of stroke
* Inability to perform study procedures
* Medical or physical conditions that would preclude participation or walking (e.g., severe arthritis or mobility problems, uncontrolled hypertension or diabetes, renal failure, history of angina with activity)
* On medications that could adversely affect cognition, eg: antipsychotics, opioids, stimulants, chemotherapy, anti-parkinsonian drugs (eg Levodopa), neurologic prescriptions to treat Multiple sclerosis and/or Parkinson's
* Psychotic disorders
* Confounding neurologic conditions (e.g., active central nervous system (CNS) opportunistic infections, seizure disorders, head injury with loss of consciousness >30 minutes, intracranial neoplasms, stroke with neurological or neuropsychiatric sequelae)
* Substance Use Disorder, Major Depressive and Generalized Anxiety Disorders within six months of evaluation

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in Adaptation Magnitude Assessed as Peak Step Length Symmetry | Baseline (Pre-training), Week 2 (Post-training)
  Locomotor adaptation is the ability to adjust stepping movements to changing environmental demands via trial-and-error processing. Step length symmetry data from the split-belt phase will be used to evaluate each individual's locomotor adaptation magnitude capacity by assessing the peak step length symmetry in the early adaptation period.
Change in Adaptation Rate Assessed as the Number of Steps to Reach Step Symmetry | Baseline (Pre-training), Week 2 (Post-training)
  The adaptation rate is assessed as the number of steps required to reach a plateau in step symmetry during late adaptation.
Change in 10-Meter Overground Walk Test | Baseline (Pre-training), Week 2 (Post-training)
  Gait speed is assessed with the 10-Meter Overground Walk Test. The 10-Meter Overground Walk Test is used to assess walking speed over a short distance. A 10 meter (m) walkway over solid flooring will be measured and marked at start (0 m), 2 m, 8 m, and finish (10 m). Participants will be asked to complete three trials of the 10 m walk at their comfortable self-selected walking speed. The time for the three trials for each speed will be averaged and gait speed converted to meters/second.
Change in 6-Minute Walk Test | Baseline (Pre-training), Week 2 (Post-training)
  Gait endurance is assessed with the 6-minute walk test. The 6-Minute Walk Test is a sub-maximal exercise test used to assess walking endurance. A walkway of a minimum 12 m over solid flooring will be measured and marked with a turn-around marked at either end of the walkway. The turn-around points will be approximately 49 inches (124 cm) wide with clear markings. A chair will be placed at one end of the walkway to allow for seated rest breaks if necessary. Prior to administering the test, the participant will be seated in the chair resting. The participant will then be asked to walk as far as possible in 6 minutes along the walkway using scripted instruction (see below). The distance (in meters) will be calculated by multiplying the number of total laps by 12 meters and adding the distance of the partial lap completed at the time the test ended.
Change in Montreal Cognitive Assessment (MoCA) Score | Baseline (Pre-training), Week 2 (Post-training)
  MoCA is an instrument to screen for mild cognitive dysfunction, assessing the cognitive domains of attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation. Total scores range from 0 to 30 with higher scores indicating better cognitive function. A normal score is considered to be 26 or higher.
Change in NIH-EXAMINER n-back Task Accuracy | Baseline (Pre-training), Week 2 (Post-training)
  The NIH-EXAMINER assesses spatial working memory with the n-back tasks. The 1-back involves maintaining and updating one location at a time while two locations at a time are maintained and updated with the 2-back. During the n-back tasks, participants view a series of stimuli and press a button when a particular stimulus has been previously shown. The 1-back consists of one block of 30 trials, ten of which match the location of the previous square, and 20 that are in a different location. The 2-back consists of one block of 90 trials, 30 of which match the location of the square two before, and 60 that are in a different location. The score is calculated as the percentage of correct responses.

SECONDARY OUTCOMES:
Change in De-adaptation Magnitude Assessed as Peak Step Length Symmetry | Baseline (Pre-training), Week 2 (Post-training)
  Step length symmetry data from the split-belt phase will be used to evaluate each individual's locomotor de-adaptation magnitude capacity by assessing the peak step length symmetry after treadmill belt speeds return to normal.
Change in De-adaptation Rate Assessed as the Number of Steps to Reach Step Symmetry | Baseline (Pre-training), Week 2 (Post-training)
  The de-adaptation rate is assessed as the number of steps required to reach a plateau in step symmetry after treadmill belt speeds return to normal.
Change in Timed Up and Go (TUG) Test | Baseline (Pre-training), Week 2 (Post-training)
  The Timed Up and Go test assesses mobility, balance, walking ability, and fall risk in older adults. The participant will be asked to be seated in a standard height chair (seat height 46 cm, arm height 67 cm), placing his/her back against the chair and resting his/her arms on the chair's arms. The participant will be asked to get up from the chair, walk to a line 3 m from the edge of the chair, turn around at the line, walk back to the chair, and sit down. The test will be timed using a stopwatch from when the investigator says "Go" to when the participant's buttocks touches the chair upon return. Time of the test will be recorded for single and dual-task conditions.
Change in Falls History | Baseline (Pre-training), Week 2 (Post-training)
  Falls incidence and risk is assessed as self-reported history of falls.
Change in Stride Duration | Baseline (Pre-training), Week 2 (Post-training)
  Gait performance is assessed as gait cycle duration, which is the time in milliseconds (ms) for the same foot to contact the floor in consecutive footsteps.
Change in Double-support Duration | Baseline (Pre-training), Week 2 (Post-training)
  Gait performance is assessed as double-support duration. Double-support is the time when both feet are contacting the ground and it increases as walking speed decreases.
Change in Executive Index Score (EIS) | Baseline (Pre-training), Week 2 (Post-training)
  Cognition is assessed with the Executive Index Score (EIS) which is based on performance on Trail-Making Test Part B, Clock Drawing, Digit Span, Letter A Tapping, Serial 7 Subtraction, Letter Fluency and Abstraction items. The EIS is calculated by adding raw scores for the included tasks. Total scores range from 0 to 13 and higher scores indicate better cognitive function.
Change in Trail Making Test Part B Score | Baseline (Pre-training), Week 2 (Post-training)
  In Part A of the Trail Making Test (TMT) participants are presented with a sheet of paper with 25 circles numbered 1 through 25. Participants are asked to draw lines connecting the circles in ascending order of the numbers. The task is scored as the amount of time it takes in seconds for the circles to be correctly connected. The average time to complete the task is 29 seconds. Times greater than 78 seconds indicate cognitive impairment.
Change in Step Length | Baseline (Pre-training), Week 2 (Post-training)
  Gait performance is assessed with step length. Step length is the distance between heel of one foot to the heel print of the other foot, measured in feet.
Change in Step Length Variability | Baseline (Pre-training), Week 2 (Post-training)
  Gait performance is assessed with the variability of step length.

CONTACTS AND LOCATIONS:
Overall Officials: Trisha Kesar, PT, PhD, Principal Investigator — Emory University
Locations (1):
- Emory Rehabilitation Hospital, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified demographic, clinical measures of walking and sensorimotor function, walking biomechanics, and electromyography (EMG) data that is collected during this study will be made available for sharing with the research community. All preprocessed data will be deposited to Distributed Archives for Neurophysiology Data Integration (DANDI) after the conclusion of the award period for this study.
Supporting Information: Analytic Code
Time Frame: The research community will have access to the data when the award for this study ends and findings from this study are published. The data will be preserved indefinitely and is subject to decisions by DANDI regarding how long data will be preserved.
Access Criteria: The research community will have unrestricted access to the data with an account through DANDI.